CLINICAL TRIAL: NCT07266402
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Parallel-Group Study of Barzolvolimab in Participants With Cold Induced Urticaria and Symptomatic Dermographism (EMBARQ-COLDU and SD)
Brief Title: A Study to Investigate Efficacy, Safety and Tolerability of Barzolvolimab Versus Placebo in Adults With Cold Induced Urticaria and Symptomatic Dermographism Inadequately Controlled by H1-antihistamines (EMBARQ - ColdU and SD)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDX0159-16
Record Dates: First submitted 2025-11-19; First posted 2025-12-05 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Chronic Inducible Urticaria; Cold Urticaria; Cold-Induced Urticaria; Symptomatic Dermographism
Keywords: Chronic Inducible urticaria; cold urticaria; cold-induced urticaria; ColdU; symptomatic dermographism,; SD; barzolvolimab; CDX0159; CDX-0159
MeSH Terms: conditions — Chronic Inducible Urticaria; Cold Urticaria; Familial dermographism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- barzolvolimab 450mg loading dose followed by 150mg in patients with Cold Induced Urticaria (Experimental): barzolvolimab 450mg injection subcutaneously at randomization , then 150mg injection subcutaneously every 4 weeks for 24 weeks
  Interventions: Drug: Barzolvolimab
- Placebo comparator in patients with Cold Induced Urticaria (Placebo Comparator): Placebo injection subcutaneously every 4 weeks for 24 weeks
  Interventions: Drug: Matching Placebo
- barzolvolimab 450mg loading dose followed by 150mg in patients with Symptomatic Dermographism (Experimental): barzolvolimab 450mg injection subcutaneously at randomization, then 150mg injection subcutaneously every 4 weeks for 24 weeks
  Interventions: Drug: Barzolvolimab
- Placebo comparator in patients with Symptomatic Dermographism (Placebo Comparator): Placebo injection subcutaneously every 4 weeks for 24 weeks
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Barzolvolimab — Subcutaneous Administration
  Other Names: CDX-0159
  Arms: barzolvolimab 450mg loading dose followed by 150mg in patients with Cold Induced Urticaria; barzolvolimab 450mg loading dose followed by 150mg in patients with Symptomatic Dermographism
Drug: Matching Placebo — Subcutaneous Administration
  Arms: Placebo comparator in patients with Cold Induced Urticaria; Placebo comparator in patients with Symptomatic Dermographism

SUMMARY:
The purpose of this Phase 3, randomized, double-blind, placebo-controlled study is to assess the activity and safety of barzolvolimab compared to placebo in participants with cold induced urticaria or symptomatic dermographism who remain symptomatic despite the use of H1-antihistamines.

DETAILED DESCRIPTION:
The purpose of this Phase 3, randomized, double-blind, placebo-controlled study is to assess the activity and safety of barzolvolimab compared to placebo in participants with cold induced urticaria (ColdU) or symptomatic dermographism (SD) who remain symptomatic despite the use of H1-antihistamines.

There is a Screening Period of up to 4 weeks, followed by a 24-week treatment period where patients will receive barzolvolimab or placebo. Patients receiving barzolvolimab will receive 450mg at the start of the treatment period and then 150mg. Then there is 16-week follow-up period where all patients are observed.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males and females, >/= 18 years of age.
2. Diagnosis of cold induced urticaria or symptomatic dermographism >/= 3 months.
3. Diagnosis of cold induced urticaria or symptomatic dermographism despite the use of a stable regimen of second generation non-sedating H1-antihistamine as defined by:

   1. The presence of hives for >/= 6 weeks at any time prior to Visit 1 despite the use of H1-antihistamines.
   2. Must be on a stable regimen of second generation non-sedating H1-antihistamine for >/= 4 weeks prior to study treatment.
   3. Cold induced urticaria: A Critical Threshold Temperature (CTT) of ≥ 10 °C and < 37 °C using the TempTest® and a numerical rating scale score of ≥ 3 for itch after the provocation test.
   4. Symptomatic dermographism: A Critical Friction Threshold (CFT) of ≥ 3 using the FricTest® and a numerical rating scale score of ≥ 3 for itch after the provocation test.
4. Cold induced urticaria: Positive ice-cube test resulting in hives at the provocation site during Screening
5. Normal blood counts and liver function tests.
6. Both males and females of child-bearing potential must agree to use highly effective contraceptives during the study and for 150 days after treatment.
7. Willing and able to complete a daily symptom electronic diary and comply with study visits.
8. Participants with and without prior biologic experience are eligible.

Key Exclusion Criteria:

1. Women who are pregnant or nursing.
2. Clearly defined cause for chronic urticaria.
3. Active, pruritic skin condition in addition to cold induced urticaria or symptomatic dermographism.
4. Medical condition that would cause additional risk or interfere with study procedures.
5. Known HIV, hepatitis B or hepatitis C infection.
6. Vaccination of a live vaccine within 2 months prior to study treatment (subjects must agree to avoid vaccination during the study). Inactivated vaccines are allowed such as seasonal influenza injection or COVID-19 vaccine.
7. History of anaphylaxis, unless due to cold exposure over a large part of the body (such as swimming in cold water).
8. Prior treatment with barzolvolimab

There are additional criteria that your study doctor will review with you to confirm you are eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Complete response to provocation testing at Week 12 | From Day 1 (first dose) to Week 12
  Proportion of Cold Induced Urticaria [ColdU] participants with complete response in Critical Temperature Threshold (CTT) or proportion of Symptomatic Dermographism [SD] participants with complete response in Critical Friction Threshold at Week 12.
  * For ColdU patients, a complete response is defined as absence of wheals at the provocation site within 10 min at ≤ 4°C after provocation using TempTest®
  * For SD patients, a complete response test is defined as absence of wheals at the provocation site within 10 min at 0 pins after provocation using the FricTest®

SECONDARY OUTCOMES:
Change from baseline in Critical Temperature Threshold (CTT) at Week 12 | From Day 1 (first dose) to Week 12
  For participants with Cold Induced Urticaria, change from baseline in CTT following the TempTest® at Week 12.
  CTT is defined as threshold temperature at which wheals are triggered (highest temperature for cold), assessed at the 10-minute mark.
Change from baseline in Critical Friction Threshold (CFT) at Week 12 | From Day 1 (first dose) to Week 12
  For participants with Symptomatic Dermographism, change from baseline in CFT following the FricTest® at Week 12.
  CFT is the threshold pin number at which wheals are triggered, assessed at the 10-minute mark.
Complete response to provocation testing at Week 24 for Cold Induced Urticaria participants | From Day 1 (first dose) to Week 24
  Proportion of Cold Induced Urticaria participants with complete response in Critical Temperature Threshold (CTT) following the TempTest® 4.0 at Week 24.
Complete response to provocation testing at Week 24 for Symptomatic Dermographism participants | From Day 1 (first dose) to Week 24
  Proportion of Symptomatic Dermographism participants with complete response in Critical Friction Threshold (CFT) following the FricTest® 4.0 at Week 24
Change from baseline in Critical Temperature Threshold (CTT) at Week 24 | From Day 1 (first dose) to Week 24
  For participants with Cold Induced Urticaria, change from baseline in CTT following the TempTest® at Week 24.
Change from baseline in Critical Friction Threshold (CFT) at Week 24 | From Day 1 (first dose) to Week 24
  For participants with Symptomatic Dermographism, change from baseline in CFT following the FricTest® at Week 24.
Improvement in clinical symptoms of itch at Week 12 | From Day 1 (first dose) to Week 12
  Change from baseline in worst itch-numerical rating scale (WI-NRS) at Week 12 (on a scale of 0-10 in which no itch/burning/pain = 0 and worst ever is = 10).
Improvement in clinical symptoms of itch at Week 24 | From Day 1 (first dose) to Week 24
  Change from baseline in worst itch-numerical rating scale (WI-NRS) at Week 24 (on a scale of 0-10 in which no itch/burning/pain = 0 and worst ever is = 10).
Change from baseline in WI-NRS following provocation testing (WI-NRSprovo) at Week 12 | From Day 1 (first dose) to Week 12
  Change from baseline in WI-NRSprovo at Week 12 (on a scale of 0-10 in which no itch/burning/pain = 0 and worst ever is = 10).
Complete response to provocation testing at Week 4 | From Day 1 (first dose) to Week 4
  Proportion of Cold Induced Urticaria participants with complete response in Critical Temperature Threshold (CTT) following the TempTest® 4.0 at Week 4 or proportion of Symptomatic Dermographism participants with complete response in Critical Friction Threshold (CFT) following the FricTest® 4.0 at Week 4
Change from baseline in Critical Temperature Threshold (CTT) at Week 4 | From Day 1 (first dose) to Week 4
  For participants with Cold Induced Urticaria, change from baseline in CTT following the TempTest® at Week 4.
Change from baseline in Critical Friction Threshold (CFT) at Week 4 | From Day 1 (first dose) to Week 4
  For participants with Symptomatic Dermographism, change from baseline in CFT following the FricTest® at Week 4.
Improvement in clinical symptoms of hives at Week 12 | From Day 1 (first dose) to Week 12
  Change from baseline in worst hives-numerical rating scale (WH-NRS) at Week 12 (on a scale of 0-10 in which no itch/burning/pain = 0 and worst ever is = 10).
Improvement in clinical symptoms of hives at Week 24 | From Day 1 (first dose) to Week 24
  Change from baseline in worst hives-numerical rating scale (WH-NRS) at Week 24 (on a scale of 0-10 in which no itch/burning/pain = 0 and worst ever is = 10).
Improvement in Dermatology Quality of Life Index (DLQI) at Week 12 | From Day 1 (first dose) to Week 12
  Proportion of participants with DLQI = 0-1 at Week 12.
Incidence of Treatment-Emergent Adverse Events | From Day 1 (first dose) to Week 40
  Occurrence of treatment emergent adverse events, adverse events of special interest and serious adverse events during the study.

CONTACTS AND LOCATIONS:
Locations (72):
- United States (26):
  - Cahaba Dermatology & Skin Health Center, LLC, Birmingham, Alabama
  - One of a Kind Clinical Research Center, LLC, Scottsdale, Arizona
  - Kern Research, Inc., Bakersfield, California
  - One of a Kind Clinical Research Center, Napa, California
  - Allergy & Asthma Consultants, Redwood City, California
  - Amicis Research Center, Sherman Oaks, California
  - FOMAT - Allergy, Asthma & Immunology Medical Group, Ventura, California
  - Direct Helpers Research Center, Hialeah, Florida
  - Well Pharma Medical Research, Corp., Miami, Florida
  - Deluxe Health Center, LLC, Miami Lakes, Florida
  - GCP, Global Clinical Professionals, St. Petersburg, Florida
  - Advanced Clinical Research Institute, Tampa, Florida
  - Centricity Research Columbus Dermatology, Columbus, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Endeavor Health Clinical Trials Center, Skokie, Illinois
  - Equity Medical, LLC, Bowling Green, Kentucky
  - Advanced ENT and Allergy, PLLC, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Revival Research Institute, LLC, Troy, Michigan
  - Equity Medical, LLC, New York, New York
  - Markowitz Medical PLLC dba OptiSkin Medical, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Advanced Dermatology and Cosmetic Surgery - Spartanburg, Spartanburg, South Carolina
  - RFSA Dermatology, San Antonio, Texas
  - Allergy Associates of Utah, Sandy City, Utah
- Germany (14):
  - Universitätsklinikum Augsburg - III. Med. Klinik, Augsburg
  - Institut für Allergieforschung (IFA) Charité - Universitätsmedizin Berlin, Berlin
  - Elbekliniken Buxtehude, Buxtehude
  - Rosenpark Research, Darmstadt
  - University Hospital Dresden, Dresden
  - University Hospital Düsseldorf, Düsseldorf
  - Universitatsklinkum Erlangen-Ulmenweg 18, Erlangen
  - Universitätsklinikum Göttingen, Göttingen
  - Universitätsklinikum Heidelberg, Heidelberg
  - MVZ DermaKiel GmbH, Kiel
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck
  - LMU Klinikum der Universität, München
  - Universitätsklinikum Münster, Klinik u. Poliklinik f. Dermatologie, Münster
  - Universitäts-Hautklinik Tübingen, Tübingen
- Lithuania (5):
  - CD8 Klinika, Kaunas
  - UAB Ausros Medicinos Centras, Kaunas
  - Republic Klaipeda Hospital, Klaipėda
  - Center of Allergy Diagnosis and Treatment, Vilnius
  - Santaros KTC (klinikiniu tyrimu centras), Vilnius
- Poland (13):
  - Centrum Medyczne ALL-MED Badania Kliniczne, Krakow
  - Centrum Nowoczesnych Terapii Dobry Lekarz Sp. z o.o., Krakow
  - "Oddzial Kliniczny Chorob Wewnetrznych, Astmy i Alergii z Odcinkiem dla Dzieci, Uniwersytecki Szpital Kliniczny nr 1 w Lodzi", Lodz
  - Santa Familia PTG Lodz, Lodz
  - Luxderm Specjalistyczny Gabinet Dermatologiczny Prof. dr hab. N. med. Dorota Krasowska, Lublin
  - Uniwersytecki Szpital Kliniczny w Opolu, Opole
  - Medicome Sp. z o.o., Oświęcim
  - EMC Instytut Medyczny S.A.PL CERTUS Szpital i Ambulatorium, Poznan
  - Uniwersytecki Szpital Kliniczny im. Fryderyka Chopina w Rzeszowie, Rzeszów
  - Alergo-med Ośrodek Badań Klinicznych Spólka z ograniczoną odpowiedzialnością, Tarnów
  - MICS Centrum Medyczne Toruń, Torun
  - Klinika Ambroziak Dermatologia, Warsaw
  - Cityclinic Przychodnia Lekarsko-Psychologiczna Matusiak Sp. Partnerska, Wroclaw
- South Africa (9):
  - Worthwhile Clinical Trials, Benoni
  - Allergy and Immunology Unit, University of Cape Town Lung Institute (UCTLI), Cape Town
  - Dr. PJ Sebastian, Durban
  - Infinity Dermatology Inc, Durban
  - Synapta Clinical Research Centre, Durban
  - Newtown Clinical Research Centre, Johannesburg
  - Sandton Medical Research Centre, Johannesburg
  - Global Clinical Trials (Pty) Ltd, Pretoria
  - Allergy and Asthma Centre, Westville
- Spain (2):
  - Hospital del Mar, Barcelona
  - Clinica Universidad Navarra - Pamplona, Pamplona
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge
  - Queen Elizabeth University Hospital, Glasgow
  - Salford Care Organisation NCA NHS Trust, Manchester